CLINICAL TRIAL: NCT01438281
Title: Phase I Study to Evaluate the Ocular Tolerance of SYL1001 in Healthy Volunteers
Brief Title: Study to Evaluate the Ocular Tolerance of SYL1001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SYL1001_I; 2010-023113-56 (EudraCT Number)
Record Dates: First submitted 2011-09-14; First posted 2011-09-22 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Ocular Pain; Dry Eye
Keywords: ocular pain; dry eye; siRNA
MeSH Terms: conditions — Eye Pain; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- SYL1001 (Experimental)
  Interventions: Drug: SYL1001

INTERVENTIONS:
Drug: SYL1001 — SYL1001 eye drops. topical administration

SUMMARY:
The purpose of this study is to determine whether SYL1001 is safe for the prevention and treatment of ocular pain and dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide signed inform consent prior to participation.
* BMI between 19,5 y 29 kg/m2.
* Normal ocular test in both eyes: IOP </=21 mmHg. BCVAof >/=0,8 (20/25)Snellen scale, or </=0.1 LogMar.
* Normal fluorescein Clearance Test in both eyes.
* Normal funduscopy in both eyes.

Exclusion Criteria:

* Pregnant or breastfeeding females or those with a positive pregnancy test or who will not use a medically acceptable contraceptive method from selection and during the study.
* Current relevant disease.
* Previous chronic processes or with rebound characteristics that could interfere with study according investigator's judgment.
* Volunteers who have received pharmacological treatment, including medicinal plants, during the four weeks previous to beginning the study.
* Having used corticoids sporadically in the last 30 days whichever the route aof administration, or any med by ocular or nasal administration route.
* Case history of hypersensitivity to meds or any other allergic process.
* Visual alterations: previous eye surgery, glaucoma, use of lenses, uveitis or ocular surface pathology (dry eye, blepharitis).
* Volunteers with visual alteration with more than 3 dioptres in either eye.
* Volunteers who has participated in a clinical trial during the past fout months before study entry.
* Blood or derivate transfusion during the six previous months to study entry.
* Case history of drug or alcohol abuse or dependence.
* Positive result in test drug abuse during selection period.
* positive serology results to hepatitis B virus(HbsAg), virus C o VIH.
* Analytic alterations medically relevant, at investigator's judgement.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Local tolerance assessment of cornea and conjunctival sac after administration of one dose of SYL1001 for period 1 and after 7 days of administration of SYL1001 with one dose per day for period 2. | Period I: 3 days, Period II: 11 days
  Local tolerance and ocular surface (cornea and conjunctival) on the area of administration 24 hours after last administration. It will be performed using a slit lamp which will be performed before, during and after the administration at established times. Adverse events will be registered and the determination of subjective tolerance will use the visual analogical scale in cases where asubjects refers them

SECONDARY OUTCOMES:
General tolerance assessment after administration of one dose of SYL1001 (period 1) and after 7 days administration (period 2) | Period I: 3 days; Period II: 11 days
  Corneal pachymetry eye exploration BCVA (best corrected visual acuity) eye fundus evaluation Clinical exploration Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Belen Sadaba, MD, PhD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Benitez-Del-Castillo JM, Moreno-Montanes J, Jimenez-Alfaro I, Munoz-Negrete FJ, Turman K, Palumaa K, Sadaba B, Gonzalez MV, Ruz V, Vargas B, Paneda C, Martinez T, Bleau AM, Jimenez AI. Safety and Efficacy Clinical Trials for SYL1001, a Novel Short Interfering RNA for the Treatment of Dry Eye Disease. Invest Ophthalmol Vis Sci. 2016 Nov 1;57(14):6447-6454. doi: 10.1167/iovs.16-20303. PMID 27893109